CLINICAL TRIAL: NCT04306445
Title: The Effect of a Gas-filled Intragastric Balloon or Endoscopic Sleeve Gastroplasty for Weight Loss Compared With a Meal Replacement Weight Loss Program on Gastric Emptying, Hormonal Adaptation to Weight Loss, and Hunger
Brief Title: How Gas-Filled Intragastric Balloons or Endoscopic Sleeve Gastroplasty Affect Hunger, Hunger Hormones, and Gastric Emptying Compared to Meal Replacements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0278
Record Dates: First submitted 2020-03-06; First posted 2020-03-13 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- GF-IGB: Obalon Balloon (Active Comparator): Obalon balloons are gas-filled balloons used for weight loss by taking up more space in the stomach. There are three separate balloons that are placed. They are inflated once the capsules containing the balloons are swallowed. The second balloon is swallowed two weeks after the first balloon, and the third balloon is swallowed four to eight weeks after the second balloon. All three balloons are removed six months after the first balloon is placed.
  Interventions: Device: GF-IGB: Obalon Balloon
- Medically Supervised Meal Replacement Program: My New Weigh (Active Comparator): Meal Replacements are used for weight loss in order to achieve a very low-calorie diet that is nutritionally balanced. Four to five meal replacements are consumed per day. If only four meal replacements are consumed per day, three servings of vegetables and two servings of fruit are consumed as well. This program lasts for about five months or twenty weeks.
  Interventions: Dietary Supplement: Medically Supervised Meal Replacement Program: My New Weigh
- Endoscopic Sleeve Gastroplasty: ESG (Active Comparator): Endoscopic sleeve gastroplasty (ESG) is a weight loss procedure that uses an endoscopic suturing device known as Overstitch to reduce the size of the stomach. This decreases the amount of food one can consume, which leads to the consumption of fewer calories throughout the day, resulting in weight loss.
  Interventions: Procedure: Endoscopic sleeve gastroplasty: (ESG)

INTERVENTIONS:
Device: GF-IGB: Obalon Balloon — The balloon, which is attached to a thin catheter, is swallowed by the patient in a standing position. Once the two-step verification of balloon passage into the stomach by both fluoroscopy and pressure reading, the balloon is inflated to a volume of 250 ml with a nitrogen-mix gas, additional imaging of the inflated balloon is obtained, the catheter is ejected from the balloon, and the catheter is pulled out through the patient's mouth. The process is repeated at week 2 for the second balloon and between weeks 4-8 for the third balloon. All patients are given an individualized calorie prescription by a registered dietitian for a goal of up to 2 pounds of weight loss per week. The balloons are removed endoscopically 6 months after placement of the first balloon. Patients also attend monthly virtual individual diet coaching and monthly virtual group behavior coaching sessions both delivered by a registered dietitian for twelve months focused on long-term behavior change.
  Arms: GF-IGB: Obalon Balloon
Dietary Supplement: Medically Supervised Meal Replacement Program: My New Weigh — Patients are given an individualized calorie prescription by a registered dietitian for a goal of 2 pounds weight loss per week. Patients are seen in a group-based program once a week focused on long-term behavior change and use meal replacements for a nutritionally balanced very low-calorie diet for 20 weeks. 4-5 meal replacements are consumed per day. If only 4 meal replacements are consumed, individuals eat 3 servings of vegetables and 2 servings of fruit per day as well.
  Arms: Medically Supervised Meal Replacement Program: My New Weigh
Procedure: Endoscopic sleeve gastroplasty: (ESG) — Endoscopic sleeve gastroplasty is a weight loss procedure that uses an FDA 510K cleared endoscopic suturing device known as Overstitch to reduce the size of the gastric body. The procedure is completed with an endoscope. It is inserted through the mouth, down the esophagus, and into the stomach. Sutures with 8-10 bites 1.5-2 cm apart in a U-shape pattern are placed starting distally 6 cm proximal to the pylorus. Additional sutures are placed moving proximally up to 2 cm distal to the gastroesophageal junction. An additional row of sutures is then placed again in the distal to proximal stomach to complete the gastroplasty. All patients are given an individualized calorie prescription by a registered dietitian for a goal of up to 2 pounds of weight loss per week. Patients also attend monthly virtual individual diet coaching and monthly virtual group behavior coaching sessions both delivered by a registered dietitian for twelve months focused on long-term behavior change.
  Arms: Endoscopic Sleeve Gastroplasty: ESG

SUMMARY:
The disease obesity continues to be a major health issue in the US with over one third of the population having a mass index >30 kg/m2. Obesity is associated with serious cardiometabolic complications including diabetes, hypertension, dyslipidemia and myocardial infarction. Rates of successful obesity treatment with weight loss and weight maintenance remain low. Several endoscopic bariatric therapies and procedures have been approved for use in the United States, including three intragastric balloon systems (2 fluid-filled and one gas-filled) and endoscopic sleeve gastroplasty (ESG), both of which have lower risks than bariatric surgery and do not alter gastrointestinal anatomy. Weight loss with all intragastric balloons and ESG is higher than lifestyle therapy or weight loss medications, but less than bariatric surgery. Unlike weight loss medications where weight loss from the medication is regained within 6-8 months after therapy ends, weight loss maintenance with intragastric balloons remains high with 66-88.5% of the weight loss maintained 6 months after device removal. Data suggests that space occupying devices with a volume of 400 ml or more in the stomach increase feelings of fullness and result in weight loss, but this does not explain the prolonged effect of weight loss maintenance after balloon removal. Although few studies have investigated the mechanism of action of fluid-filled balloons and one study with 4 patients undergoing ESG on weight loss, these data suggest that gastric emptying as well as space occupation contribute to weight loss. However, no studies have investigated the mechanisms of action of gas filled intragastric balloons on weight loss.

Understanding the mechanisms responsible for weight loss with the gas filled intragastric balloon system and ESG as well as any weight loss independent effects on blood glucose control would lay the groundwork for studies evaluating predictors of response to improve patient selection as well as studies understanding the mechanisms behind weight loss maintenance and developing strategies to prolong weight loss maintenance.

Therefore, the purpose of this pilot study is to determine the effects 10% total body weight loss (%TBWL) in patients with obesity treated with the intragastric balloon (GF- IGB) system or ESG compared to patients with obesity treated with a meal replacement program (MRP) on 1) gastric emptying, 2) hormonal adaptation to weight loss and 3) hunger.

DETAILED DESCRIPTION:
Obesity is a chronic disease, which is associated with and contributes to multiple medical co- morbidities including but not limited to cardiovascular disease, diabetes, nonalcoholic fatty liver disease, and many different cancers. Obesity is also associated with an increased risk of all-cause mortality. Despite these known risks, treatment remains limited. This has contributed to the increase in the prevalence of obesity with 42.4%% of adults in the US adults having a body mass index (BMI) >30 kg/m2.

Endoscopic bariatric therapies are a new class of treatment for obesity, which have demonstrated more weight loss than lifestyle therapy alone and fewer complications than bariatric surgery with less weight loss than bariatric surgery. Four endoscopic devices are currently approved by the FDA for the treatment of obesity, including two intragastric balloons (IGB). One of the balloons systems are fluid filled (FF-IGB) and one is gas filled (GF-IGB). Although the GF-IGB system is swallowed, all the balloon systems require an endoscopist for endoscopic removal. In clinical registry series, these balloons demonstrate similar weight loss at 6 months. Unlike weight loss medications, weight loss maintenance is prolonged after IGB removal, which was demonstrated meta-analysis of studies and case series outside of the US of the single FF-IGB demonstrated weight loss maintenance after balloon removal 9 and in the US pivotal trials. While the occupancy of space in the stomach by IGB is known to induce satiation and satiety, this mechanism is only present with the IGB in place. Therefore, the prolonged effects of weight loss maintenance after IGB removal suggest other mechanisms contributing to weight loss with IGB treatment beyond space occupation. ESG is completed endoscopically with a device that has FDA 510k clearance for tissue apposition in the GI tract. Weight loss with ESG in a recent meta-analysis in 1772 patients demonstrated 16.5% TBWL at 12 months and 17.2% TBWL at 18-245 months. Understanding the mechanisms contributing to weight loss with the GF-IGB system and ESG will lay the groundwork for future studies to enhance the effect of IGBs and ESG on initial weight loss, patient selection, and weight loss maintenance; increasing benefits to patients treated with IGBs or ESG.

FF-IGB are known to delay gastric emptying. This is consistent with practice patterns as patients reliably have food left in their stomachs after an overnight fast requiring multiple days of liquid diet prior to endoscopic removal to avoid aspiration. In one study, the FF-IGB delayed gastric emptying compared to both baseline and a control group and the change in gastric emptying was associated with weight loss. Gastric emptying has been studied in only 4 patients before and after ESG. In these 4 patients, there was a 90-minute increase to the time for 50% of emptying of solid foods, however the limited number of patients in that study reduce overall certainty of the effect of ESG on gastric emptying. No studies have investigated the effects of the GF-IGB on gastric emptying. This protocol will clarify the effects of the GF-IGB and ESG on gastric emptying compared with a control group matched on weight loss. This will elucidate the weight loss independent effects of the devices since patients will be studied at baseline and 10% total body weight loss.

Another possible mechanism by which IGBs and ESG may induce weight loss and weight loss maintenance is through alterations in gut hormones. Ghrelin is a hormone secreted by X/A like cells, which are predominantly in the fundus of the stomach. Ghrelin concentrations fluctuate with eating, increasing pre-meals and decreasing in response to food in the stomach. Moreover, infusion of ghrelin stimulates eating in humans and is the only known hormone secreted from the GI tract to stimulate hunger. Weight loss with lifestyle therapy alone has been shown to increase fasting and meal test "active" or acyl-ghrelin concentrations, which correlated with increased hunger on visual analogue scale (VAS) testing. Acyl-Ghrelin concentrations were still elevated at one year after weight loss despite weight regain of almost 50%, which suggests that acyl-ghrelin plays and important role in weight regain. Studies investigating ghrelin concentrations in the setting of FF-IGBs have been mixed, demonstrating decreased fasting plasma total ghrelin concentrations, no change in fasting or meal test ghrelin concentrations in FF-IGB or control groups, increased fasting plasma ghrelin compared to a control group at months 1 and 6 with decreased ghrelin in the active arm compared to the control arm after removal and increased ghrelin concentrations in a single arm. However, these studies measured total ghrelin not acyl ghrelin. This limits the reliability of the data especially since no change in ghrelin concentrations were seen in control patients with weight loss in which an increase in acyl- ghrelin is expected. Moreover, all the studies were with FF-IGB and none were in the GF-IGB system.

Balloon type may have an effect on acyl-ghrelin concentrations, as GF-IGB tend to float in the fundus and body of the stomach, which may affect the IGB's ability to suppress acyl-ghrelin secretion. In one of the aforementioned studies a post-hoc analysis demonstrated that the small number of patients whose FF-IGBs localized to the fundus had greater suppression of ghrelin.

Fasting ghrelin has been evaluated in one study with 12 patients pre and post ESG. Fasting ghrelin concentrations did not increase with weight loss, but meal testing was not performed.

Therefore, this protocol will determine the effects of 10% TBWL from either GF-IGB system treatment or ESG treatment compared to lifestyle and meal replacement therapy on acyl-ghrelin concentrations, the active form of ghrelin, which stimulates hunger, and the sensation of hunger with the VAS. This will allow for the detection of effects that are specific to either procedure and independent of weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 22-65
* Weight Stable (<5% weight change in the last 3 months)
* Initiating treatment with GF-IGB, ESG, or medically supervised MRP
* BMI of 30-40

Exclusion Criteria:

* History of liver disease
* History of uncontrolled thyroid disease
* History of anemia
* History of diabetes
* History of eating disorder
* History of uncontrolled depression defined as a score of ≥ 10 on PHQ-9 (Patient Health Questionnaire-9)
* Use of weight loss medications in the past 3 months
* History of gastroparesis
* History of bariatric surgery
* History to allergy or intolerance to any component of the meal used in the gastric emptying study or mixed meal test
* Women who are pregnant or lactating
* Currently incarcerated
* Non English speaking
* Decisionally challenged adults

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2024-03-02 (Estimated); Study Completion 2024-03-02 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 6 months
  10%TBWL by GI-IGB, ESG, or Medically Supervised MRP

SECONDARY OUTCOMES:
Gastric emptying measured by technetium 99 gastric emptying study | 6 months
  The investigators hypothesize that treatment with GF-IGB and ESG will result in greater gastric retention of contents at 2 hours compared with patients who are treated with MRP.
Acyl-Ghrelin measured at multiple times points during a mixed meal test (MMT) | 6 months
  The investigators hypothesize that weight loss induced increase in active ghrelin concentrations seen during a mixed meal tolerance test will be lower in patients treated with GF- IGB and ESG compared with patients treated with MRP.
Glucose measured at multiple times points during a mixed meal test (MMT) | 6 months
  There will be no difference in glucose concentrations in patients treated with GF-IGB and ESG compared with treatments treated with MRP.
Insulin measured at multiple times points during a mixed meal test (MMT) | 6 months
  There will be no difference in insulin concentrations in patients treated with GF-IGB and ESG compared with treatments treated with MRP.
Level of hunger measured using a visual analog scale (Hunger VAS) | 6 months
  The investigators hypothesize that hunger will increase before and during a MMT after weight loss with MRP but will not change from baseline after weight loss with GF-IGB and ESG treatment. Scales will range from 0-100, with 100 being more hungry (worse outcome) and 0 being less hungry (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Sullivan, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Courcoulas A, Abu Dayyeh BK, Eaton L, Robinson J, Woodman G, Fusco M, Shayani V, Billy H, Pambianco D, Gostout C. Intragastric balloon as an adjunct to lifestyle intervention: a randomized controlled trial. Int J Obes (Lond). 2017 Mar;41(3):427-433. doi: 10.1038/ijo.2016.229. Epub 2016 Dec 23. PMID 28017964
- [Background] Ponce J, Woodman G, Swain J, Wilson E, English W, Ikramuddin S, Bour E, Edmundowicz S, Snyder B, Soto F, Sullivan S, Holcomb R, Lehmann J; REDUCE Pivotal Trial Investigators. The REDUCE pivotal trial: a prospective, randomized controlled pivotal trial of a dual intragastric balloon for the treatment of obesity. Surg Obes Relat Dis. 2015 Jul-Aug;11(4):874-81. doi: 10.1016/j.soard.2014.12.006. Epub 2014 Dec 16. PMID 25868829
- [Background] Thompson CC, Abu Dayyeh BK, Kushner R, Sullivan S, Schorr AB, Amaro A, Apovian CM, Fullum T, Zarrinpar A, Jensen MD, Stein AC, Edmundowicz S, Kahaleh M, Ryou M, Bohning JM, Ginsberg G, Huang C, Tran DD, Glaser JP, Martin JA, Jaffe DL, Farraye FA, Ho SB, Kumar N, Harakal D, Young M, Thomas CE, Shukla AP, Ryan MB, Haas M, Goldsmith H, McCrea J, Aronne LJ. Percutaneous Gastrostomy Device for the Treatment of Class II and Class III Obesity: Results of a Randomized Controlled Trial. Am J Gastroenterol. 2017 Mar;112(3):447-457. doi: 10.1038/ajg.2016.500. Epub 2016 Dec 6. PMID 27922026
- [Background] Sullivan S, Swain J, Woodman G, Edmundowicz S, Hassanein T, Shayani V, Fang JC, Noar M, Eid G, English WJ, Tariq N, Larsen M, Jonnalagadda SS, Riff DS, Ponce J, Early D, Volckmann E, Ibele AR, Spann MD, Krishnan K, Bucobo JC, Pryor A. Randomized sham-controlled trial of the 6-month swallowable gas-filled intragastric balloon system for weight loss. Surg Obes Relat Dis. 2018 Dec;14(12):1876-1889. doi: 10.1016/j.soard.2018.09.486. Epub 2018 Sep 29. PMID 30545596
- [Background] Agnihotri A, Xie A, Bartalos C, Kushnir V, Sullivan S, Islam S, Islam E, Lamet M, Lamet A, Farboudmanesch R, Overholt BF, Altawil J, Early DS, Bennett M, Lowe A, Mullady DK, Adeyeri CS, El Zein M, Mishra P, Fayad L, Dunlap M, Oberbach A, Cheskin LJ, Kalloo AN, Khashab MA, Kumbhari V. Real-World Safety and Efficacy of Fluid-Filled Dual Intragastric Balloon for Weight Loss. Clin Gastroenterol Hepatol. 2018 Jul;16(7):1081-1088.e1. doi: 10.1016/j.cgh.2018.02.026. Epub 2018 Mar 2. PMID 29481969
- [Background] Vargas EJ, Pesta CM, Bali A, Ibegbu E, Bazerbachi F, Moore RL, Kumbhari V, Sharaiha RZ, Curry TW, DosSantos G, Schmitz R, Agnihotri A, Novikov AA, Pitt T, Dunlap MK, Herr A, Aronne L, Ledonne E, Kadouh HC, Cheskin LJ, Mundi MS, Acosta A, Gostout CJ, Abu Dayyeh BK. Single Fluid-Filled Intragastric Balloon Safe and Effective for Inducing Weight Loss in a Real-World Population. Clin Gastroenterol Hepatol. 2018 Jul;16(7):1073-1080.e1. doi: 10.1016/j.cgh.2018.01.046. Epub 2018 Feb 7. PMID 29425781
- [Background] Geliebter A, Westreich S, Gage D. Gastric distention by balloon and test-meal intake in obese and lean subjects. Am J Clin Nutr. 1988 Sep;48(3):592-4. doi: 10.1093/ajcn/48.3.592. PMID 3414573
- [Background] Gomez V, Woodman G, Abu Dayyeh BK. Delayed gastric emptying as a proposed mechanism of action during intragastric balloon therapy: Results of a prospective study. Obesity (Silver Spring). 2016 Sep;24(9):1849-53. doi: 10.1002/oby.21555. Epub 2016 Jul 28. PMID 27465076
- [Background] Mion F, Napoleon B, Roman S, Malvoisin E, Trepo F, Pujol B, Lefort C, Bory RM. Effects of intragastric balloon on gastric emptying and plasma ghrelin levels in non-morbid obese patients. Obes Surg. 2005 Apr;15(4):510-6. doi: 10.1381/0960892053723411. PMID 15946431
- [Background] Ariyasu H, Takaya K, Tagami T, Ogawa Y, Hosoda K, Akamizu T, Suda M, Koh T, Natsui K, Toyooka S, Shirakami G, Usui T, Shimatsu A, Doi K, Hosoda H, Kojima M, Kangawa K, Nakao K. Stomach is a major source of circulating ghrelin, and feeding state determines plasma ghrelin-like immunoreactivity levels in humans. J Clin Endocrinol Metab. 2001 Oct;86(10):4753-8. doi: 10.1210/jcem.86.10.7885. PMID 11600536
- [Background] Wren AM, Seal LJ, Cohen MA, Brynes AE, Frost GS, Murphy KG, Dhillo WS, Ghatei MA, Bloom SR. Ghrelin enhances appetite and increases food intake in humans. J Clin Endocrinol Metab. 2001 Dec;86(12):5992. doi: 10.1210/jcem.86.12.8111. PMID 11739476
- [Background] Sumithran P, Prendergast LA, Delbridge E, Purcell K, Shulkes A, Kriketos A, Proietto J. Long-term persistence of hormonal adaptations to weight loss. N Engl J Med. 2011 Oct 27;365(17):1597-604. doi: 10.1056/NEJMoa1105816. PMID 22029981
- [Background] Martinez-Brocca MA, Belda O, Parejo J, Jimenez L, del Valle A, Pereira JL, Garcia-Pesquera F, Astorga R, Leal-Cerro A, Garcia-Luna PP. Intragastric balloon-induced satiety is not mediated by modification in fasting or postprandial plasma ghrelin levels in morbid obesity. Obes Surg. 2007 May;17(5):649-57. doi: 10.1007/s11695-007-9109-z. PMID 17658025
- [Background] Mathus-Vliegen EM, Eichenberger RI. Fasting and meal-suppressed ghrelin levels before and after intragastric balloons and balloon-induced weight loss. Obes Surg. 2014 Jan;24(1):85-94. doi: 10.1007/s11695-013-1053-5. PMID 23918282
- [Background] Konopko-Zubrzycka M, Baniukiewicz A, Wroblewski E, Kowalska I, Zarzycki W, Gorska M, Dabrowski A. The effect of intragastric balloon on plasma ghrelin, leptin, and adiponectin levels in patients with morbid obesity. J Clin Endocrinol Metab. 2009 May;94(5):1644-9. doi: 10.1210/jc.2008-1083. Epub 2009 Mar 3. PMID 19258408
- [Background] Buzga M, Evzen M, Pavel K, Tomas K, Vladislava Z, Pavel Z, Svagera Z. Effects of the intragastric balloon MedSil on weight loss, fat tissue, lipid metabolism, and hormones involved in energy balance. Obes Surg. 2014 Jun;24(6):909-15. doi: 10.1007/s11695-014-1191-4. PMID 24488758
- [Background] Sullivan S, Kirk EP, Mittendorfer B, Patterson BW, Klein S. Randomized trial of exercise effect on intrahepatic triglyceride content and lipid kinetics in nonalcoholic fatty liver disease. Hepatology. 2012 Jun;55(6):1738-45. doi: 10.1002/hep.25548. Epub 2012 Apr 25. PMID 22213436
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Yanovski SZ, Marcus MD, Wadden TA, Walsh BT. The Questionnaire on Eating and Weight Patterns-5: an updated screening instrument for binge eating disorder. Int J Eat Disord. 2015 Apr;48(3):259-61. doi: 10.1002/eat.22372. Epub 2014 Dec 26. No abstract available. PMID 25545458
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity and Severe Obesity Among Adults: United States, 2017-2018. NCHS Data Brief. 2020 Feb;(360):1-8. PMID 32487284
- [Background] Moore RL, Seger MV, Garber SM, Smith AB, Nguyen RT, Shieh MK, Snow RG, Sullivan S. Clinical safety and effectiveness of a swallowable gas-filled intragastric balloon system for weight loss: consecutively treated patients in the initial year of U.S. commercialization. Surg Obes Relat Dis. 2019 Mar;15(3):417-423. doi: 10.1016/j.soard.2018.12.007. Epub 2018 Dec 6. PMID 30797717
- [Background] ASGE Bariatric Endoscopy Task Force and ASGE Technology Committee; Abu Dayyeh BK, Kumar N, Edmundowicz SA, Jonnalagadda S, Larsen M, Sullivan S, Thompson CC, Banerjee S. ASGE Bariatric Endoscopy Task Force systematic review and meta-analysis assessing the ASGE PIVI thresholds for adopting endoscopic bariatric therapies. Gastrointest Endosc. 2015 Sep;82(3):425-38.e5. doi: 10.1016/j.gie.2015.03.1964. Epub 2015 Jul 29. PMID 26232362
- [Background] Hedjoudje A, Abu Dayyeh BK, Cheskin LJ, Adam A, Neto MG, Badurdeen D, Morales JG, Sartoretto A, Nava GL, Vargas E, Sui Z, Fayad L, Farha J, Khashab MA, Kalloo AN, Alqahtani AR, Thompson CC, Kumbhari V. Efficacy and Safety of Endoscopic Sleeve Gastroplasty: A Systematic Review and Meta-Analysis. Clin Gastroenterol Hepatol. 2020 May;18(5):1043-1053.e4. doi: 10.1016/j.cgh.2019.08.022. Epub 2019 Aug 20. PMID 31442601
- [Background] Abu Dayyeh BK, Acosta A, Camilleri M, Mundi MS, Rajan E, Topazian MD, Gostout CJ. Endoscopic Sleeve Gastroplasty Alters Gastric Physiology and Induces Loss of Body Weight in Obese Individuals. Clin Gastroenterol Hepatol. 2017 Jan;15(1):37-43.e1. doi: 10.1016/j.cgh.2015.12.030. Epub 2015 Dec 31. PMID 26748219
- [Background] Lopez-Nava G, Negi A, Bautista-Castano I, Rubio MA, Asokkumar R. Gut and Metabolic Hormones Changes After Endoscopic Sleeve Gastroplasty (ESG) Vs. Laparoscopic Sleeve Gastrectomy (LSG). Obes Surg. 2020 Jul;30(7):2642-2651. doi: 10.1007/s11695-020-04541-0. PMID 32193741
- [Background] Wilson EB, Noren E, Gruvaeus J, Paradis C. A comparative 100-participant 5-year study of aspiration therapy versus Roux-en-Y gastric bypass: 2nd and 3rd year results. Surgery for Obesity and Related Diseases 2018; 14(11):S15.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04306445/Prot_SAP_002.pdf
  • Informed Consent Form (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT04306445/ICF_003.pdf